CLINICAL TRIAL: NCT03123497
Title: Assessment of Quality of Life of Children With Chronic Idiopathic Thrombocytopenic Purpura
Brief Title: Assessment of Quality of Life of Children With Chronic Idiopathic Thrombocytopenic Purpura (Kid's ITP Tools)
Acronym: KIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC17_0011
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idiopathic Thrombocytopenic Purpura: completion of questionnaire
  Interventions: Other: completion of questionnaire

INTERVENTIONS:
Other: completion of questionnaire — completion of questionnaire for patient and parent

SUMMARY:
Assessment of quality of life of patient with chronic idiopathic thrombocytopenic purpura according to the type of treatment

ELIGIBILITY:
Inclusion Criteria:

* children with Idiopathic thrombocytopenic purpura
* aged between 1 and 17 year
* Idiopathic thrombocytopenic purpura persistent at 12 months
* obtention of informed consent

Exclusion Criteria:

* Persistant/acute Idiopathic thrombocytopenic purpura
* concomittant chronic disease, stabilized or not
* Concomittant disease with life expectancy < 1 year
* Person who have not belong to a social security scheme
* Secondary Idiopathic thrombocytopenic purpura

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with idiopathic thombocytopenic purpura, aged between 1 and 17 year
Sampling Method: Non-Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
quality of life score according to type of treatment | at inclusion visit
  quality of life score according to type of treatment

SECONDARY OUTCOMES:
number of hospitalisation and consults per year | at inclusion visit
  number of hospitalisation and consults per year
description of general quality of life | at inclusion visit
  use ped'sQL general
description of general quality of life | at inclusion visit
  use ped'sQL fatigue
description of awareness of parent and patient about Idiopathic thrombocytopenic purpura | at inclusion visit
  use Kid's ITO Tools questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Pellier, Pr, Principal Investigator — chu
Locations (1):
- CHU d'Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No